CLINICAL TRIAL: NCT00731237
Title: XIENCE V® Everolimus Eluting Coronary Stent System (EECSS) EXCEED: Evaluation of XIENCE V® Catheterization Lab Endpoints and Excellence in Delivery
Brief Title: XIENCE V® EXCEED: Evaluation of XIENCE V® Catheterization Lab Endpoints and Excellence in Delivery
Acronym: EXCEED
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Matt Kiely, Manager Medical Information, Abbott Vascular
Other Study IDs: 08-382
Record Dates: First submitted 2008-08-05; First posted 2008-08-08 (Estimated); Last update posted 2009-10-16 (Estimated); Status verified 2009-10

CONDITIONS: Atherosclerosis; Coronary Artery Disease
Keywords: Drug Eluting Stent; Percutaneous Coronary Intervention; Everolimus
MeSH Terms: conditions — Atherosclerosis; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: The procedures undergone by this group will be evaluated for: Acute performance, deliverability and resource utilization during the procedure in the catheterization lab during commercial use by various physicians with a range of coronary stenting experience.

SUMMARY:
This trial is to assess physician-determined XIENCE V® EECSS acute performance, deliverability and resource utilization in the catheterization lab during commercial use by various physicians with a range of coronary stenting experience

DETAILED DESCRIPTION:
This study will evaluate overall physician-determined XIENCE V® Everolimus Eluting Coronary Stent system (XIENCE V®) acute performance, deliverability and resource utilization in the catheterization lab in the "real world" as used by a broad group of physicians at a variety of health care facilities. This study will include all consecutively enrolled patients in the United States of America (USA) who consent to participate and receive XIENCE V® stents.

ELIGIBILITY:
General Inclusion Criteria:

* The patient agrees to participate in this study by signing the IRB approved informed consent form prior to the index procedure.
* Alternatively, the patient's legally authorized representative agrees to the patient's participation in this study and signs the informed consent form prior to the index procedure.

General Exclusion Criteria:

* Inability to obtain an informed consent is an exclusion criterion.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients undergoing planned or possible PCI should be invited to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 2517 (Actual)
Dates: Start 2008-10; Primary Completion 2009-03 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Overall physician-determined XIENCE V® EECSS acute performance and deliverability. | acute
Physician-determined procedure success | acute

SECONDARY OUTCOMES:
Individual component of adjunctive devices and drugs used during procedure. Number and type of guide wires | acute
Individual component of adjunctive devices and drugs used during procedure. Number and type of guiding catheters | acute
Individual component of adjunctive devices and drugs used during procedure. Number and type of balloon dilation catheters | acute
Individual component of adjunctive devices and drugs used during procedure: Balloon pressures (pre-dilation/post-dilation pressures) | acute
Individual component of adjunctive devices and drugs used during procedure: Number of stents | acute
Individual component of adjunctive devices and drugs used during procedure: Amount of radiographic contrast | acute
Individual component of adjunctive devices and drugs used during procedure: Fluoroscopy time | acute
Individual component of adjunctive devices and drugs used during procedure: Duration of PCI procedure | acute
Individual component of adjunctive devices and drugs used during procedure: IVUS use | acute
Individual component of adjunctive devices and drugs used during procedure: Thienopyridine loading dose (prior to, during or after procedure) | acute
Individual component of adjunctive devices and drugs used during procedure: Aspirin loading dose (prior to, during or after procedure) | acute
Device Success | acute

CONTACTS AND LOCATIONS:
Overall Officials: John McPherson, MD, Principal Investigator — Vanderbuilt University
Locations (44):
- United States (44):
  - The Heart Center, PC, Huntsville, Alabama
  - Arizona Regional Medical Center, Mesa, Arizona
  - Tri Lakes Research-Central Arkansas Cardiovascular, Hot Springs, Arkansas
  - Tri Lakes Research-Central Arkansas Cardiovascular, Hot Springs Village, Arkansas
  - NEA Baptist Memorial Hospital, Jonesboro, Arkansas
  - La Mesa Cardiac Center, La Mesa, California
  - Pikes Peak Cardiology, Colorado Springs, Colorado
  - University of Connecticut Health Center, Farmington, Connecticut
  - Bradenton Heart Research Center, Bradenton, Florida
  - Ocala Regional Medical Center, Ocala, Florida
  - Harbin Clinic LLC, Rome, Georgia
  - Sherman Hospital, Elgin, Illinois
  - Heart Care Research Foundation, Mokena, Illinois
  - Northern Indiana Research Alliance, Fort Wayne, Indiana
  - Clarian Health Partners - Methodist Hospital, Indianapolis, Indiana
  - Medical Consultants PC, Muncie, Indiana
  - Iowa Heart Center, Des Moines, Iowa
  - University of Iowa Hospital, Iowa City, Iowa
  - Promise Regional Medical Center - Hutchinson, Hutchinson, Kansas
  - Allegiance Health, Jackson, Michigan
  - Michigan Cardiovascular Institute, Midland, Michigan
  - Michigan Cardio Vascular Institute at St. Mary's of MI, Saginaw, Michigan
  - Coast Cardiovascular Consultants, P.L.L.C, Biloxi, Mississippi
  - St. Luke's, Kansas City, Missouri
  - St. Johns Mercy Medical Center, St Louis, Missouri
  - Renown Regional Medical Center, Reno, Nevada
  - AtlantiCare Regional Medical Center, Pomona, New Jersey
  - University of New Mexico Health Sciences Center, Albuquerque, New Mexico
  - First Health Moore Regional Hospital, Pinehurst, North Carolina
  - Fairfield Cardiac Cath Lab, LLC, Fairfield, Ohio
  - Smith Clinic, Marion, Ohio
  - St. Anthony Hospital, Oklahoma City, Oklahoma
  - Conemaugh Valley Memorial Hospital, Johnstown, Pennsylvania
  - The Good Samaritan Hospital, Lebanon, Pennsylvania
  - Phoenixville Hospital, Phoenixville, Pennsylvania
  - University Pittsburgh Medical Center (UPMC), Pittsburgh, Pennsylvania
  - UPMC Presbyterian Shadyside Hospital, Pittsburgh, Pennsylvania
  - Palmetto Health Clinic, Columbia, South Carolina
  - Piedmont Medical Center / Carolina Cardiology Associates, Rock Hill, South Carolina
  - Wellmont Bristol Regional Medical Center, Bristol, Tennessee
  - Tomball Regional Medical Center, Tomball, Texas
  - Virginia Cardiovascular Specialists, Richmond, Virginia
  - Cardiovascular Associates, Ltd., Virginia Beach, Virginia
  - CAMC Health Education and Research Institute, Inc., Charleston, West Virginia